CLINICAL TRIAL: NCT04472481
Title: Vitamin D: Does It Help Tregs in Active Rheumatoid Arthritis Patients.
Brief Title: Vitamin D Effect in Rheumatoid Arthritis.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Souzan Ezzat Gado, Lecturer of Rheumatology,physical medicine &Rehabilitation., Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 33846
Record Dates: First submitted 2020-07-07; First posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Active Rheumatoid Arthritis
Keywords: Regulatory T cell; Foxp3+; vitamin D supplementation; Rheumatoid arthritis; DMARD
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Ergocalciferols; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- group II (Other): 50000 IU of Vitamin D2 (Ergocalciferol 1.25 mg tablet) weekly for 3 months
  Interventions: Drug: Ergocalciferol 1.25 mg tablet

INTERVENTIONS:
Drug: Ergocalciferol 1.25 mg tablet — weekly 50000 IU of Vitamin D2 (Ergocalciferol 1.25 mg tablet) given orally group II

SUMMARY:
Regulatory T (Tregs) cells play an important role in the maintenance of immunological tolerance. It decrease in the peripheral blood of rheumatoid arthritis patients. Vitamin D has an immunomodulatory and anti-inflammatory effect in rheumatoid arthritis.

Vitamin D supplementation significantly enhances Tregs percentage in the peripheral blood of RA patients. So supplementation of Vit D improves rheumatoid arthritis disease activity.

DETAILED DESCRIPTION:
Background: Regulatory T cells (Tregs) play an important role in the maintenance of immunological tolerance, so Tregs deficiency or decrease suppressor functions may be associated with development of autoimmune diseases.

Vitamin D is essential for normal bone mineralization and growth, prevention of osteopenia, osteoporosis, and nonspecific painful musculoskeletal conditions . Vitamin D is thought to have an immunomodulatory and anti-inflammatory actions, as its receptors are widely expressed in peripheral mononuclear blood cells, also its deficiency associated with several autoimmune disorders, including rheumatoid arthritis

Methods: 40 patients with active RA were randomly assigned into two groups. Group I received MTX plus hydroxychloroquine, group II received MTX and hydroxychloroquine plus vitamin D supplementation for 3 months, in addition to 30 healthy volunteers as control group. Peripheral blood Tregs were measured by Flow Cytometry.

Statistical Analysis. The collected data analyzed by SPSS software (version 16). The range, mean and standard deviation were calculated for quantitative variables. Categorical variables were expressed as number and percentages; Chi square was used as a test of their significance. Skewness, kurtosis; Shapiro-Wilk, and The Kolmogorov-Smirnov tests were used to test the normality for the data. The difference between two means was analyzed using the students (t) test (paired and unpaired samples- T tests). Significance was considered at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* disease duration less than 3 years from the time of diagnosis, age more than 18 years, a diagnosis of RA according to the 2010 ACR/ EULAR Classification criteria for RA diagnosis , active disease according to DAS-28, for those receiving nonsteroidal anti-inflammatory drugs and corticosteroids, the dosage had to be stable for at least 2 weeks before screening.

Exclusion Criteria:

* Patients with allergic, and infectious diseases, patients receiving steroids for the first time within 2 weeks before the study, patients with hypercalcemia, hypercalciuria, nephrolithiasis, or neoplastic diseases were excluded from the study. We also excluded patients on any biologic therapy and patients with prior use of leflunomide, hydroxychloroquine, or sulphasalazine for more than 2 months.

Ages: 33 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2019-12-22 (Actual); Study Completion 2020-03-22 (Actual)

PRIMARY OUTCOMES:
change from base line Measurement of regulatory T cells (CD4+CD25+FoxP3+) at 3 months | base line and after 3 months
  4 ml of heparinized blood from the subjects' peripheral blood was collected. Human peripheral blood natural regulatory T cells (Tregs) were surface stained with Mouse Anti-Human CD4 FITC (Fluorescein) conjugated Monoclonal Antibody and Mouse Anti-Human IL-2 Rα/CD25 APC (allophycocyanin) conjugated Monoclonal Antibody, followed by intracellular staining using Rabbit Anti-Human/ Mouse FoxP3 PE (phycoerythrin) conjugated Antigen Affinity-purified Monoclonal Antibody, cells were fixed and permeabilized with FoxP3 Fixation & Permeabilization Buffer Kit. Cells were gated on lymphocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Souzan E Gado, MD, Principal Investigator — Lecturer; Hanaa S EL-banna, MD, Principal Investigator — Lecturer
Locations (1):
- Souzan Ezzat Gado, Tanta, EL-gharbia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Z, Chang C, Lu Q. Epigenetics of CD4+ T cells in autoimmune diseases. Curr Opin Rheumatol. 2017 Jul;29(4):361-368. doi: 10.1097/BOR.0000000000000393. PMID 28362657
- [Background] Lan Q, Fan H, Quesniaux V, Ryffel B, Liu Z, Zheng SG. Induced Foxp3(+) regulatory T cells: a potential new weapon to treat autoimmune and inflammatory diseases? J Mol Cell Biol. 2012 Feb;4(1):22-8. doi: 10.1093/jmcb/mjr039. Epub 2011 Nov 22. PMID 22107826
- [Derived] El-Banna HS, Gado SE. Vitamin D: does it help Tregs in active rheumatoid arthritis patients. Expert Rev Clin Immunol. 2020 Aug;16(8):847-853. doi: 10.1080/1744666X.2020.1805317. Epub 2020 Aug 25. PMID 32783547